CLINICAL TRIAL: NCT06738823
Title: Effect of Wii Fit Training in Comparison to Vestibular Rehabilitation Training on Balance in Patients With Benign Paroxysmal Postional Vertigo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/52
Record Dates: First submitted 2024-11-28; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Benign Paroxysmal Positional Vertigo; Balance; Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): The participants will receive intervention through Wii fit training which includes games tight rope tension, ski slalom, penguin slide, table tilt, and heading for 6 total 6 weeks.
  3 days per week session will be given for 30 minutes including 5-minutes warmup and cool down and 5 minutes of break in between to avoid fatigue.
  Interventions: Procedure: INTERVENTION GROUP : TRAINING WITH WIIFIT
- Experimental group B (Active Comparator): The participants will receive vestibular rehabilitation training. The rehabilitation programme will include weight shifting, neck rotations, sit to stand exercises on padded mat, and head movements with eyes closed.
  The intervention will be given for 3 minutes, 3 days a week for total 6 weeks of time period.
  Interventions: Procedure: VESTIBULAR REHABILITATION TRAINING

INTERVENTIONS:
Procedure: INTERVENTION GROUP : TRAINING WITH WIIFIT — RCT (RANDOMIZED CONTROL TRIAL) GROUP 1 : Wii FIT TRAINING TIGHT ROPE TENSION, SKI SLALOM, PENGUIN SLIDE, TABLE TILT GROUP 2 : VESTIBULAR REHABILITATION TRAINING WEIGHT SHIFTING, NECK ROTATIONS, SIT TO STAND EXERCISES ON PADDED MAT AND HEAD MOVEMENTS WITH EYES CLOSED.
  Arms: Experimental group A
Procedure: VESTIBULAR REHABILITATION TRAINING — WEIGHT SHIFTING, NECK ROTATIONS, SIT TO STAND EXERCISES ON PADDED MAT AND HEAD MOVEMENTS WITH EYES CLOSED.
  Arms: Experimental group B

SUMMARY:
THIS STUDY IS A RANDOMIZED CONTROL TRIAL AND THE PURPOSE OF THE STUDY IS TO DETERMINE THE EFFECT OF WIIFIT TRAINING IN COMPARISON TO VESTIBULAR REHAB TRAINING ON BALANCE IN PATIENTS WITH BENIGN PAROXYSMAL POSITIONAL VERTIGO

DETAILED DESCRIPTION:
Effects of wiifit training will be assessed for balance and vertigo which includes the parameters of balance training.

Benign Paroxysmal Positional Vertigo patients aged 30-60 years The participants will be assessed through Vestibular Rehabilitation questionnaire (VRBQ), Dizziness handicap inventory (DHI), Functional reach test, Clinical test for sensory integration in balance and vertigo symptom scale.

Informed consent will be taken after which the participants will be recruited into two groups, where one group will receive wiifit training and other group will receive vestibular rehabilitation training.

Base-line and post-treatment measurement will be taken for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with benign paroxysmal positional vertigo.
* Aged 30-60 years.
* Ability to stand and walk independently.
* Male and Female
* Positive Dix Hallpike Test
* DHI Scale: 36-42 (moderate Handicap)

Exclusion Criteria:

* patients with history of vestibular surgery or cochlear implantation.
* Patients with history of seizures or epilepsy.
* patients with a pacemaker or implantable cardioverter-defibrillator(ICD).
* Patients with history of severe head injury or concussion within the past year.
* No other vestibular disorders or conditions that may affect balance.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Static Balance | 6 weeks
  The Vestibular Rehabilitation Benefit Questionnaire (VRBQ) is a validated tool used to measure balance 0 means no problem, 100 means severe problem
Vertigo | 6 weeks
  DHI scale is used to assess vertigo.The questionnaire consists of 25 items with 3 responses YES= 4 points SOMETIMES = 2 points and NO = 0 points. The total score ranges from 0 to 100, higher score indicating self perceived handicap due to dizziness.
Static Balance | 6 weeks
  CTSIB of Biodex is used to assess static balance and has 4 components. a) Firm surface with eyes open; (Mean value 0.44)test the integration of visual,somatosensory and vestibular inputs. All sensory systems are available for balance. b) Firm surface with eyes closed; (mean value 0.80)evaluate the reliance on somatosensory input for balance and visual input is eliminated.c) Foam surface with eyes open; (Mean value; 0.79) Test the ability to use visual and vestibular inputs for balance when somatosensory inputs is unreliable,unstable surface. d) Foam surface with eyes closed; (mean value 2.41) primarily challenges the vestibular system by eliminating visual input and providing unreliable somatosensory feedback. The total mean of these 4 components is 1.11.
Dynamic balance | 6 weeks
  Functional Reach test will be used to assess dynamic balance
  * Scoring:
  * Distance in centimeters or inches is recorded.
  * Normal values :
  * <15 cm indicates a high fall risk in older adults

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan